CLINICAL TRIAL: NCT04904016
Title: A Single Center, Open, Non-controlled Pilot Investigation to Evaluate FLowOx2.0™ for Experimental Treatment of Spasticity With Concomitant Pain in Multiple Sclerosis, Using Intermittent Negative Pressure Affecting Arteriovenous Reflex
Brief Title: Pilot Investigation to Evaluate FlowOx2.0™ for Experimental Treatment of Spasticity
Acronym: FlowOx-MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Otivio AS (Industry)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FO-NP001_29032021
Record Dates: First submitted 2021-05-04; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Multiple Sclerosis; Spasticity, Muscle; Pain
Keywords: Blood flow; FlowOx™; Stiffness
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention FlowOx treatment (Experimental): Each participating subject will be provided with one FlowOx™ system, which will be used about 1 hour per day every day of the week for a 4-week period with the option to extend the treatment time to up to 6 months if the patients would like to continue.
  Interventions: Device: FlowOx™

INTERVENTIONS:
Device: FlowOx™ — The FlowOx™ system generates a negative oscillating pressure which cause rapid fluctuations in blood flow in the leg and foot.

SUMMARY:
This is a descriptive, prospective, non-controlled clinical investigation to be conducted on approximately 10 enrolled subjects at one site at Haukeland University Hospital in Bergen, Norway. The target subjects are male or female, 18-70 years, diagnosed with MS according to revised McDonald criteria (9) with spasticity and pain associated with the spasticity. Spasticity is evaluated based on self-reported spasticity using the numerical rating scale (NRS) which describes the average score of spasticity over the last 24 hours at >4 (where the scale scores spasticity from 0-10, where 0 is no spasticity, and 10 is worst possible spasticity), - combined with pain in the lower extremities last 24 hours. The pilot investigation is done to evaluate if FlowOx2.0™ can be used to treat spasticity with concomitant pain in patients with multiple sclerosis, using intermittent negative pressure affecting arteriovenous reflex.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnose MS according to revised McDonald criteria
2. Give written informed consent.
3. Have an age between 18-70 years.
4. Have stable disease without attack or progression of loss of function in the last three months.
5. Have self-reported spasticity, scored using the numeric rating scale (NRS) which describes the average score of spasticity over the last 24 hours, at ≥ 4 (where the scale scores spasticity from 0-10, where 0 is no spasticity, and 10 is worst possible spasticity), - combined with pain in the lower extremities last 24 hours
6. Have tried standard treatment for spasticity and pain without achieving a satisfactory effect.
7. Stable and unchanged treatment of spasticity and pain the last month
8. Stable and unchanged disease-modulating treatment for MS last 6 months.
9. Function level measured by the Expanded Disability Status Scale (EDSS) 2.0-6.5
10. Can self-manage study equipment.

Exclusion Criteria:

1. Have spasticity due to a disease other than MS.
2. Pregnancy or plan a pregnancy within the upcoming study period of 6 months.
3. Have an ongoing infection.
4. Have received botulinum toxin injection for spasticity within the last 4 months.
5. Have symptoms or illness that make it difficult to participate in the study.
6. Having planned surgery or other treatment within the coming study period of 6 months makes it difficult to participate in the study.
7. Have functional scores outside inclusion criteria measured by EDSS 2.0-6.5
8. Have had disease activity beyond requirements for stable disease as described in inclusion criteria
9. Have changed drug treatment beyond requirements for stable treatment as described in inclusion criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-05-28 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Self-Reported Spasticity, using Numerical Rating Scale: | 4 weeks
  The unabbreviated scale title: Numerical Rating Scale The minimum and maximum values: 0, 10 Higher scores mean a worse outcome.
  To evaluate change in self-reported spasticity using the numerical rating scale (NRS) over the last 24 hours after daily 1-hour self-treatment with FlowOx from baseline to week 4

SECONDARY OUTCOMES:
Desire to continue treatment | 4 weeks
  Proportion of patients who wish to continue treatment with FlowOx beyond 4 weeks
Self-Reported Spasticity, using Numerical Rating Scale | 3 months, 6 months
  The unabbreviated scale title: Numerical Rating Scale The minimum and maximum values: 0, 10 Higher scores mean a worse outcome.
  To evaluate change in self-reported spasticity using the numerical rating scale (NRS) over the last 24 hours after daily 1-hour self-treatment with FlowOx compared to baseline
Spasticity - modified Ashworth Scale | 4 weeks, 3 months and 6 months
  The unabbreviated scale title: Modified Ashworth Scale The minimum and maximum values: 0, 4 Higher scores mean a worse outcome.
  Change in spasticity measured by modified Ashworth scale from baseline to week 4, month 3 and month 6.
Self-reported pain using Numerical Rating Scale | 4 weeks, 3 months and 6 months
  The unabbreviated scale title: Numerical Rating Scale The minimum and maximum values: 0, 10 Higher score means worse pain.
  To evaluate change in self-reported spasticity using the numerical rating scale (NRS) over the last 24 hours after daily 1-hour self-treatment with FlowOx from baseline.
T25-FW | 4 weeks, 3 months, 6 months
  Change of Timed 25-Foot Walk (T25-FW) from baseline
Expanded Disability Status Scale | 4 weeks, 3 months, 6 months
  The unabbreviated scale title: Expanded Disability Status Scale The minimum and maximum values: 0, 10 Higher score means worse disability status.
  Change of functional score measured by Expanded Disability Status Scale (EDSS) and compared to baseline
Self-reported sleep (NRS) | 4 weeks, 3 months, 6 months
  The unabbreviated scale title: Numerical Rating Scale The minimum and maximum values: 0, 10 Higher score means worse sleep. Change in self reported sleep quality will measured by (NRS) and compared to baseline
Hospital Anxiety and Depression Scale | 4 weeks, 3 months, 6 months
  The unabbreviated scale title: Hospital Anxiety and Depression Scale The minimum and maximum values: 0, 3 Higher score means worse outcome. The Scale has 14 questions, the scores will be summarized at each time point and compared to baseline
Fatigue Scale for Motor and Cognitive Functions | 4 weeks, 3 months, 6 months
  The unabbreviated scale title: Fatigue Scale for Motor and Cognitive Functions (FSMC) The FSMC is an assessment of MS-related cognitive and motor fatigue. A Likert-type 5-point scale (ranging from 'does not apply at all' to 'applies completely') produces a score between 1 and 5 for each scored question. Thus minimum value is 20 (no fatigue at all) and maximum value is 100 (severest grade of fatigue). Two subscales (mental and physical fatigue) can be made. Items included in the subscale mental are 1-4-7-8-11-13-15-17-18-20 and items included in the subscale physical are 2-3-5-6-9-10-12-14-16-19. Changes in the scores will be compared to baseline.
Multiple Sclerosis Impact Scale (MSIS-29) | 4 weeks, 3 months, 6 months
  The unabbreviated scale title: Multiple Sclerosis Impact Scale The minimum and maximum values: 1, 5 Higher score means worse condition. There are 29 questions, change in reported status will be compared to baseline
SDMT | 4 weeks, 3 months, 6 months
  Change in cognition measured by the Symbol Digit Modalities Test (SDMT)
  The Symbol Digit Modalities Test (SDMT) is a cognitive task. It consists of a sheet of paper with, at the top, a sequence of nine symbols and nine corresponding numbers (key). The task sequence consists of a series of symbols, each with a blank space underneath. Within a 90-second time limit the subject is required, consulting the key as necessary, to insert the numbers associated with the symbols. Changes in the performance will be compared to baseline.
Change in medication | 4 weeks, 3 months and 6 monhts
  Medication used by the patients at the start of the trial will be recorded. Any change in frequency of use or dose of the medication to treat spasticity an/or pain will be recorded and compared to baseline.
Compliance | 4 weeks, 3 months, 6 months
  "Compliance" / use of FlowOx, is automatically logged in the machine and will be read after 4 weeks
Safety- Incidence of device related adverse and serious adverse events | 4 weeks, 3 months, 6 months
  The number and type of adverse events and servere device related events during the study will be recorded. To evaluate safety of FlowOx by assessment of device deficiencies and adverse events, non-serious and serious, rated for causality

CONTACTS AND LOCATIONS:
Overall Officials: Kjell-Morten Myhr, Principal Investigator — Neuro-SysMed, Haukeland University Hospital, Bergen Norway
Locations (1):
- Neuro-SysMed, Dept. of Neurology, Haukeland University Hospital, & Dept. of Clinical Medicine, University of Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No